CLINICAL TRIAL: NCT07064473
Title: EASi-PROTKT™ - A Phase III Double-blind, Randomised, Parallel-group Superiority Trial to Evaluate Efficacy and Safety of the Combined Use of Oral Vicadrostat (BI 690517) and Empagliflozin Compared With Placebo and Empagliflozin in Participants With Type 2 Diabetes, Hypertension and Established Cardiovascular Disease
Brief Title: EASi-PROTKT™ - A Study to Test Vicadrostat (BI 690517) Taken Together With Empagliflozin in People With Type 2 Diabetes, High Blood Pressure, and Cardiovascular Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1378-0041; U1111-1319-9064 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP)); 2025-521188-11-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Cardiovascular Diseases | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vicadrostat + empagliflozin treatment arm (Experimental)
  Interventions: Drug: Vicadrostat; Drug: Empagliflozin
- Vicadrostat-placebo + empagliflozin treatment arm (Active Comparator)
  Interventions: Drug: Empagliflozin; Drug: Placebo matching Vicadrostat

INTERVENTIONS:
Drug: Vicadrostat — Vicadrostat
  Other Names: BI 690517
  Arms: Vicadrostat + empagliflozin treatment arm
Drug: Empagliflozin — Empagliflozin
Drug: Placebo matching Vicadrostat — Placebo matching Vicadrostat
  Arms: Vicadrostat-placebo + empagliflozin treatment arm

SUMMARY:
This study is open to adults with type 2 diabetes, high blood pressure, and cardiovascular disease. People can join the study if they have these conditions and do not have a history of heart failure. The purpose of this study is to find out if a medicine called vicadrostat, when taken with empagliflozin, helps reduce cardiovascular risk in people with these conditions. The study will compare this combination to a placebo version of vicadrostat with empagliflozin.

Participants are put into 2 groups randomly, which means by chance. One group takes vicadrostat and empagliflozin tablets, and the other group takes placebo tablets with empagliflozin. Placebo tablets look like vicadrostat tablets but do not contain any medicine.

Participants take a tablet once per day for 2 and a half years and up to 4 years and 3 months. All participants also continue their medication for type 2 diabetes, high blood pressure, and cardiovascular disease. Participants have an equal chance of receiving the study medicine or placebo.

Participants are in the study for up to 4 years and 3 months. During this time, they visit the study site regularly. During these visits, doctors collect information about participants' health and take blood samples. The doctors document when participants experience cardiovascular events. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria :

* At least 18 years old at time of consent
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2).
* Participants with medical history of hypertension and on active pharmacological treatment
* Participants with medical history of type 2 diabetes mellitus (T2DM) and on active pharmacological treatment
* Established cardiovascular (CV) disease and on active pharmacological treatment
* At least one additional risk factor for developing heart failure (HF)

Exclusion Criteria:

* History of HF or hospitalization for HF or treatment of HF
* Atrial fibrillation or Atrial flutter with a resting heart rate >110 beats per minute (bpm) documented by echocardiogram (ECG) at Visit 1 (screening)
* Advanced untreated conduction disease or untreated clinically relevant ventricular arrhythmia at Visit 1 (screening)
* Treatment with an Mineralocorticoid receptor antagonist (MRA)
* Treatment with amiloride or other potassium-sparing diuretic
* Receiving the following treatments at Visit 1 (screening) or requiring such treatment before Visit 2 (randomisation), or planned during the trial:

  * A direct renin inhibitor (e.g. aliskiren)
  * More than one Angiotensin-converting enzyme inhibitor (ACEi) and/or Angiotensin receptor blocker (ARB) (including Angiotensin receptor-neprilysin inhibitor (ARNi)) used simultaneously
  * Other aldosterone synthase inhibitors (e.g. baxdrostat)
  * Systemic mineralocorticoid replacement therapy (e.g. fludrocortisone) Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11800 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2029-12-14 (Estimated); Study Completion 2029-12-21 (Estimated)

PRIMARY OUTCOMES:
Time to first event of cardiovascular (CV) death or heart failure event (HFE) | Up to 51 months

SECONDARY OUTCOMES:
Time to first event of cardiovascular (CV) death or hospitalisation for heart failure (HHF) | Up to 51 months
Absolute change from baseline in mean systolic blood pressure (SBP) [mmHg] at Week 24 | At baseline and week 24
Relative change from baseline in Urine Albumin Creatinine Ratio (UACR) [mg/g] at Week 24 | At baseline and week 24
Time to first occurrence of the composite outcome of kidney disease progression, HHF, CV death | Up to 51 months
Time to first event of CV death, HFE, non-fatal myocardial infarction (MI) or non-fatal stroke (4-point Major adverse cardiovascular events (MACE)) | Up to 51 months
Occurrences of all-cause hospitalisations (first and recurrent) | Up to 51 months
Time to first event of new-onset atrial fibrillation or atrial flutter (in participants without history of atrial fibrillation and atrial flutter) or CV death | Up to 51 months
Time to all-cause death | Up to 51 months
Time to CV death | Up to 51 months
Time to first HHF | Up to 51 months
Time to first event of new-onset HF or CV death | Up to 51 months
Occurrences of HHF (first and recurrent) | Up to 51 months
Absolute change from baseline in mean diastolic blood pressure (DBP) [mmHg] at Week 24 | At baseline and week 24

CONTACTS AND LOCATIONS:
Locations (1149):
- United States (217):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Eastern Shore Research Group, Fairhope, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Arizona Clinical Trials - Chandler, Chandler, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Sun City West, Arizona
  - Fiel Family & Sports Medicine, Tempe, Arizona
  - Arizona Clinical Trials, Tucson, Arizona
  - Yuma Clinical Trials, Yuma, Arizona
  - National Heart Institute - Beverly Hills, Beverly Hills, California
  - Hope Clinical Research, Canoga Park, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Velocity Clinical Research-Huntington Park, Huntington Park, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - ARK Clinical Research, Long Beach, California
  - Diabetes Associates Medical Group, Orange, California
  - Empire Clinical Research, Pomona, California
  - Velocity Clinical Research - San Bernardino, San Bernardino, California
  - Acclaim Clinical Research, San Diego, California
  - NorthBay Clinical Research, LLC, Santa Rosa, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Blue Coast Research Center, LLC, Vista, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - OptumCare Clinical Trials, LLC, Golden, Colorado
  - Cardiology Physicians of Fairfield County - Bridgeport, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Cardiology Associates of Fairfield County, Stamford, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - University Clinical Research Deland, LLC, DeLand, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Covenant Metabolic Specialists, LLC - Fort Myers, Fort Myers, Florida
  - Velocity Clinical Research-Hallandale Beach-67888, Hallandale, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Northeast Research Institute, Jacksonville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - East Coast Institute for Research, LLC - Southside, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Walgreens - Kissimmee - Site 4442, Kissimmee, Florida
  - East Coast Institute for Research - Lake City, Lake City, Florida
  - Clinical Research of Central Florida - Lakeland, Lakeland, Florida
  - Finlay Medical Research Corp, Miami, Florida
  - Optimus U Corporation-Miami-69452, Miami, Florida
  - Oceane7 Clinical Research, Miami, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - IMIC Inc., Miami, Florida
  - Alma Clinical Research, Inc., Miami, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Florida Institute for Clinical Research, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Center for Diabetes, Obesity and Metabolism, Pembroke Pines, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Covenant Metabolic Specialists, LLC - Brandon, Riverview, Florida
  - East Coast Institute for Research, LLC-Saint Augustine-63032, Saint Augustine, Florida
  - IMA Clinical Research St. Petersburg, St. Petersburg, Florida
  - Covenant Metabolic Specialists, LLC - Sarasota, University Park, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Centricity Research, Endocrine Consultants, Columbus, Georgia
  - NSC Research Inc, Johns Creek, Georgia
  - Physicians Research Associates, LLC, Lawrenceville, Georgia
  - The Jones Center for Diabetes and Endocrine Wellness, Macon, Georgia
  - Urban Family Practice Associates, PC, Marietta, Georgia
  - Javara-Savannah-67450, Savannah, Georgia
  - Javara Research - Thomasville, Thomasville, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Rocky Mountain Clinical Research - Idaho Falls, Idaho Falls, Idaho
  - Cedar Crosse Research Center, Chicago, Illinois
  - Walgreens - Chicago - Site 162, Chicago, Illinois
  - Accellacare of Duly - Lombard, Lombard, Illinois
  - Accellacare of Duly, Oak Lawn, Illinois
  - American Health Network - Avon, Avon, Indiana
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - American Health Network - Franklin, Franklin, Indiana
  - American Health Network - Greenfield, Greenfield, Indiana
  - American Health Network - Muncie, Muncie, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - AMR El Dorado, El Dorado, Kansas
  - Cotton O'Neil Diabetes & Endocrinology Center, Topeka, Kansas
  - Tekton Research - Wichita, Wichita, Kansas
  - Qualmedica Research - Bowling Green, Bowling Green, Kentucky
  - The Research Group of Lexington, Lexington, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Grace Research, LLC-Bossier City-51040, Bossier City, Louisiana
  - Louisiana Heart Center - Covington, Covington, Louisiana
  - IMA Clinical Research Monroe, Monroe, Louisiana
  - Grace Research, LLC-Shreveport-64616, Shreveport, Louisiana
  - Louisiana Heart Center - Slidell, Slidell, Louisiana
  - Monroe Research, LLC, West Monroe, Louisiana
  - Southern Clinical Research - Zachary, Zachary, Louisiana
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Medstar Montgomery Medical Center, Olney, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - TidalHealth, Inc., Salisbury, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Walgreens - Malden - Site 4966, Malden, Massachusetts
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Revival Research Institute, LLC - Dearborn, Dearborn, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - Elite Research Center, LLC, Flint, Michigan
  - Advanced Cardiology Associates, Rochester Hills, Michigan
  - Oakland Medical Center, Troy, Michigan
  - Prime Health and Wellness, Fayette, Mississippi
  - Memorial Hospital Gulfport, Gulfport, Mississippi
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Billings Clinic - Billings, Billings, Montana
  - Methodist Physicians Clinic, Fremont, Nebraska
  - Omaha VA Medical Center, Omaha, Nebraska
  - Quality Clinical Research - Omaha, Omaha, Nebraska
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - Walgreens - North Las Vegas - Site 5814, North Las Vegas, Nevada
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - NJ Heart LLC, Linden, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - New Mexico Clinical Research and Osteoporosis Center, Inc., Albuquerque, New Mexico
  - IMA Clinical Research Albuquerque, Albuquerque, New Mexico
  - Albany Med Health System - Washington Avenue Extension, Albany, New York
  - Velocity Clinical Research - Binghamton, Binghamton, New York
  - RCR - Buffalo, Buffalo, New York
  - NYC Research Inc., New York, New York
  - New York Cardiovascular Specialist PC, New York, New York
  - Northwell Health - Peconic Bay Medical Group at Riverhead, Riverhead, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Southgate Medical Group/ Southgate Medical Park, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - Cary Cardiology, Cary, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - IMA Clinical Research Lenoir, Lenoir, North Carolina
  - Accellacare-Mooresville-69123, Mooresville, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Accellacare-Wilmington-67123, Wilmington, North Carolina
  - Wake Forest University Health Sciences-Winston-Salem-61707, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - The Christ Hospital, Cincinnati, Ohio
  - Velocity Clinical Research-Cincinnati-69044, Cincinnati, Ohio
  - Centricity Research-Columbus-68879, Columbus, Ohio
  - Remington-Davis Clinical Research, Inc, Columbus, Ohio
  - Clinical Research Institute of Ohio, LLC, Westlake, Ohio
  - Tekton Research-Edmond-68875, Edmond, Oklahoma
  - South Oklahoma Heart Research Group, Oklahoma City, Oklahoma
  - Tekton Research-Yukon-68998, Yukon, Oklahoma
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Tristar Clinical Investigations PC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians-Pittsburgh-63932, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc, Pittsburgh, Pennsylvania
  - Frontier Clinical Research LLC - Scottdale, Scottdale, Pennsylvania
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians-Uniontown-69137, Uniontown, Pennsylvania
  - Suburban Research Associates, West Chester, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Piedmont Research Partners, LLC, Fort Mill, South Carolina
  - Velocity Clinical Research-Gaffney-69046, Gaffney, South Carolina
  - Tribe Clinical Research LLC, Greenville, South Carolina
  - Velocity Clinical Research-Union-68888, Union, South Carolina
  - Dunes Clinical Research, Dakota Dunes, South Dakota
  - Alliance for Multispecialty Research, LLC-Knoxville-69693, Knoxville, Tennessee
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - South Texas Research Institute-Brownsville-68426, Brownsville, Texas
  - Headlands Research, Brownsville, Texas
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - Javara Inc / Texas Health Care, PLLC, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - South Texas Research Institute-Edinburg-67012, Edinburg, Texas
  - Academy Of Diabetes, Thyroid And Endocrine, PA, El Paso, Texas
  - Care United Research, Forney, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Victorium Clinical Research, Houston, Texas
  - Houston Research Institute, Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes Institute, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Pinnacle Clinical Research, LLC, San Antonio, Texas
  - Tekton Research-San Antonio-68916, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Javara Inc. and Privia Medical Group Gulf Coast, PLLC, San Marcos, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Javara Inc.-Stephenville-68996, Stephenville, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Velocity Clinical Research, Waco, Waco, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Olympus Family Medicine, Salt Lake City, Utah
  - Velocity Clinical Research-West Jordan-69043, West Jordan, Utah
  - Seven Corners Medical Center, Falls Church, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - York Clinical Research, Norfolk, Virginia
  - Dominion Medical Associates - Downtown, Richmond, Virginia
  - Richmond VA Medical Center, Richmond, Virginia
  - Selma Medical Associates, Winchester, Winchester, Virginia
  - Universal Research Group, LLC, Tacoma, Washington
  - Frontier Clinical Research, LLC - Morgantown, Morgantown, West Virginia
  - Clinical Investigation Specialists, Inc.-Kenosha-69111, Kenosha, Wisconsin
  - Aspirus Research Institute, Wausau, Wisconsin
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Argentina (27):
  - CEC- Centro de Especialidades Cardiovasculares, Bahía Blanca
  - IDIM - Instituto de Diagnostico e Investigaciones Metabolicas, Buenos Aires
  - Buenos Aires Macula S.A., Buenos Aires
  - Centro Medico Fleischer, CABA
  - CPSIC SRL - Cardiologia Palermo, CABA
  - Sanatorio Anchorena, CABA
  - STAT Research, CABA
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Mautalen- Salud e Investigacion, CABA
  - Equipo Ciencia, CABA
  - Sanatorio Güemes, Capital Federal
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Centro Medico Viamonte, Ciudad Autonoma de Bs As
  - Consultorio de Investigacion Clinica EMO SRL, Ciudad Autonoma de Buenos Aire
  - Centro Diabetologico Dr Waitman, Córdoba
  - Clinica Universitaria Reina Fabiola - Universidad Catolica de Cordoba, Córdoba
  - Cemaic (Centro de Especialidades Medicas Ambulatorias E Investigacion Clinica), Córdoba
  - Instituto Privado de Investigaciones Clinica Cordoba S.A., Córdoba
  - CIPADI - Centro Integral de Prevención y Atención en Diabetes, Godoy Cruz
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Hospital Privado - Centro Medico de Cordoba S.A., Parque Velez Sarsfield
  - Instituto Medico Rio Cuarto, Río Cuarto
  - Instituto Medico Catamarca - IMEC, Rosario
  - Centro de Investigaciones Clinicas Baigorria, Santa Fe
  - CEDIR Santa Fe, Santa Fe
  - Centro de Investigaciones Clínicas del Litoral, Santa Fe
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Australia (26):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Blacktown Hospital, Blactown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Sydney Cardiometabolic Centre, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Heart of Australia, Chelmer, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Life Clinical Research, Ipswich, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Nightingale Research Pty Ltd, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Advara Heart Care-Leabrook-69072, Leabrook, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Health, Clayton, Victoria
  - The Northern Hospital, Epping, Victoria
  - Nightingale Research Victoria, Frankston, Victoria
  - Heartwest, Hoppers Crossing, Victoria
  - Cabrini Health, Malvern, Victoria
  - Advara HeartCare - Mulgrave, Mulgrave, Victoria
  - Advara Heartcare Research WA, Joondalup, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Austria (7):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - LKH Salzburg University Hospital, Salzburg
  - Wiener Gesundheitsverbund Klinik Favoriten, Vienna
  - Hospital Hietzing, Vienna
  - Herz Zentrum Währing, Vienna
  - Imed-19 privat, Vienna
  - Clinic Floridsdorf, Vienna
- Belgium (12):
  - AZORG Ziekenhuis, Aalst
  - Anima Research Center, Alken
  - Bonheiden - HOSP Imelda, Bonheiden
  - ULB Hopital Erasme, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Research Link, Gozée
  - Jessa Ziekenhuis, Hasselt
  - UZ Leuven, Leuven
  - CHR de la Citadelle, Liège
  - Meclinas, Mechelen
  - Roeselare - HOSP AZ Delta, Roeselare
- Brazil (23):
  - Centro de Pesquisa Clínica do Coração, Aracaju - SE
  - Centro de Pesquisa do Hospital Evangélico de Belo Horizonte, Belo Horizonte
  - AngioKormann Blumenau, Blumenau
  - Centro de Pesquisa Clinica do Brasil Ltda, Brasília
  - Hospital PUC-Campinas, Campinas
  - I9 Pesquisas Clinicas - Loema Instituto de Pesquisa Clínica e Consultores SS Ltda, Campinas
  - Núcleo de Pesquisa Clínica do ICBS/PUCPR, Curitiba
  - Centro de Pesquisas em Diabetes e Doencas Metabolicas, Fortaleza
  - Clínica CENDI Endocrinologia e Diabetes, Goiânia
  - Centro Multidisciplinar de Ensino Especializado e Pesquisa CMEP, Joinville
  - CESMAC - Hospital do Coração de Alagoas, Maceió
  - CPHosp Manaus, Manaus
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas - CePCLIN RN, Natal
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Hospital Mae de Deus, Porto Alegre
  - Clinicor Clínica Cardiológica LTDA/ Cardio Prime - CAPED, Ribeirão Preto
  - Instituto Brasil de Pesquisa Clinica (IBPClin), Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Irmandade da Santa Casa de Misericórdia de São Paulo - IPEC - Instituto de Pesquisa Clínica, Santa Cecília
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - Cpquali Pesquisa Clinica Ltda, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica, São Paulo
  - INCOR e Hospital das Clínicas da Universidade de São Paulo, São Paulo
- Bulgaria (17):
  - Diamedical Medical Center 2013, Dimitrovgrad
  - Multy profile hospital for active treatment Sv.Ivan Rilski, Dupnitsa
  - Medical Center New Polyclinic Gabrovo Ltd., Gabrovo
  - Medical Center Hera - Kyustendil EOOD, Kyustendil
  - Ambulatory Individual Practice for Cardiology Specialized Medical Care, Pernik
  - Ambulatory for Individual Practice for Specialized Medical Care in Cardiology - Dr Nikolay Iliev, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - MHAT "St. Caridad", Plovdiv
  - Diagnostic Consultative Centre Ascendent EOOD, Sofia
  - Medical Center For Specialized Medical Help In Cardiovascular Diseases OOD, Sofia
  - University Hospital Lozenetz, Sofia
  - Medical Center Hera EOOD, Sofia
  - ASOMHIDC - Individual practice "Cardio Tonus" EOOD, Sofia
  - Medical Center Medicabilis Ltd., Sofia
  - Medical Center Zara-Med EOOD, Stara Zagora
  - UMHAT Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
  - MHAT St Panteleimon, Yambol
- Canada (34):
  - CaRe Clinic (Calgary), Calgary, Alberta
  - CARe Clinic (Red Deer), Red Deer, Alberta
  - Medical Arts Research (Kelowna), Kelowna, British Columbia
  - Fraser Clinical Trials, New Westminster, British Columbia
  - Medical Arts Research (North Vancouver), North Vancouver, British Columbia
  - Medical Arts Research (Penticton), Penticton, British Columbia
  - SMH Cardiology Clinical Trials Inc., Surrey, British Columbia
  - GA Research Associates Ltd., Moncton, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Saul Vizel Medicine Professional Corporation, Cambridge, Ontario
  - Medical Trust Clinics, Courtice, Ontario
  - Centre for Studies in Family Medicine, Western University (LHRI), London, Ontario
  - KMH Cardiology Centres (Mississauga), Mississauga, Ontario
  - PACE (Partners in Advanced Cardiac Evaluation), Newmarket, Ontario
  - James Cha, MD, Oshawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - CardioQuest Research Centre, Sarnia, Ontario
  - Heart Health Institute (Scarborough), Scarborough Village, Ontario
  - KMH Cardiology Centers (Hamilton), Stoney Creek, Ontario
  - Stouffville Medical Research Institute Inc., Stouffville, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - ViaCar Recherches Cliniques Inc. (Greenfield Park), Greenfield Park, Quebec
  - Diex Recherche (Joliette), Joliette, Quebec
  - THEO Medical - Concorde (Laval), Laval, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Endocrinologie Oasis Inc, Montreal, Quebec
  - Centre de Medecine Metabolique de Lanaudiere, Terrebonne, Quebec
  - Diex Recherche (Trois-Rivieres), Trois-Rivières, Quebec
  - Diex Recherche (Quebec), Québec
- Chile (6):
  - Centros Médicos Espacio Eme SpA, Ñuñoa
  - Servicios Medicos Godoy Limitada, Providencia
  - Centro UC Investigación Clinica CICUC, Santiago
  - Smolam P.R.O, Santiago
  - Sociedad Medica Cardiologica El Llano, Santiago
  - CINVEC - Centro de Investigacion Clinica V Reg.,Vina del Mar, Viña del Mar
- China (62):
  - Baotou Central Hospital, Baotou
  - China-Japan Friendship Hospital, Beijing
  - Xuanwu Hospital,Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Province People's Hospital, Changchun
  - China-Japan Union Hospital of Jilin University, Changchun
  - Changsha Central Hospital, Changsha
  - The Second Xiangya Hospital Of Central South University, Changsha
  - The third xiangya hospital of Central South University, Changsha
  - The Third Hospital of Changsha, Changsha
  - Changzhou Second People's Hospital, Changzhou
  - West China Hospital, Sichuan University, Chengdu
  - People's Hospital of Sichuan Province, Chengdu
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Center Hospital of Dalian, Dalian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - NanFang Hosptial, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Hainan General Hospital, Haikou
  - Zhejiang Province People's Hospital, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - Forth Clinical Hospital of Harbin Medical University, Harbin
  - Anhui Provincial Hospital, Hefei
  - Huizhou Central People's Hospital, Huizhou
  - Center Hospital of Jinan, Jinan
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou
  - Lanzhou University Second Hospital, Lanzhou
  - Lishui Municipal Central Hospital, Lishui
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Luoyang Third People's Hospital, Luoyang
  - University Hospital_Macau University of Science and Technology, Macau
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Nanchang People's Hospital, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The People's Hospital Of Guangxi Zhuang Autonomous Region, Nanning
  - Affiliated Hospital of Nantong University, Nantong
  - Nanyang Second General Hospital, Nanyang
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Pingxiang People's Hospital, Pingxiang
  - First Hospital of Qinhuangdao, Qinhuangdao
  - Centre Hospital of Putuo District, Shanghai, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - People's Hospital of Liaoning Province, Shenyang
  - Siping Central People's Hospital, Siping
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Union Medical Center Nankai University Affiliated Hospital, Tianjin
  - The Fourth Central Hospital of Tianjin, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Hubei Province Zhongshan Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Shaanxi Provincial People's Hospital, Xi'an
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen
  - Xiangyang Central Hospital, Xiangyang
  - Xianyang Hospital of Yan'an University, Xianyang
  - The People's Hospital Of Xuancheng City, Xuancheng
  - Affiliated Hospital, Xuzhou Medical college, Xuzhou
  - General Hospital of Ningxia Medical University, Yinchuan
  - Affiliated Hospital of Jiangsu University, Zhenjiang
  - Zibo Municipal Hospital, Zibo
- Colombia (9):
  - Cardiomet CEQUIN S.A.S, Armenia
  - Clínica de la Costa SAS, Barranquilla
  - IPS Centro Cientifico-Asistencial S.A.S, Barranquilla
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Corazon IPS S.A.S., Barranquilla
  - IPS médicos internistas de Caldas S.A.S., Manizales
  - Rodrigo Botero S.A.S., Medellín
  - Hospital Pablo Tobón Uribe, Medellín
  - Cardiomet Pereira, Pereira
- Croatia (7):
  - International Medical Center Priora, Čepin
  - Special Hospital for Medical Rehabilitation Krapinske Toplice, Krapinske Toplice
  - Thalassotherapy Opatija, Opatija
  - Polyclinic Slavonija, Osijek, Osijek
  - Specialty Hospital Medico, Rijeka
  - Poliklinika Bonifarm Zagreb, Zagreb
  - Solmed Polyclinic, Zagreb
- Czechia (11):
  - Medicus Services Ltd., Brandýs nad Labem
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Kardiologická ambulance Brno s.r.o, Brno
  - Vojenska nemocnice Brno, Brno
  - DIKa centrum s.r.o., Havířov
  - Kardiologie a angiologie s.r.o, Prague
  - Endokrinologicky ustav, Prague
  - University Thomayer´s Hospital, Prague
  - MILAN KVAPIL s.r.o., Prague
  - Clinical Trials Services s.r.o, Uherské Hradiště
  - KIGE s.r.o., Znojmo
- Denmark (8):
  - Aarhus University Hospital, Aarhus N
  - Esbjerg Sygehus, Esbjerg
  - Herlev and Gentofte Hospital, Herlev
  - Steno Diabetes Center Copenhagen, Herlev
  - Regionshospitalet Gødstrup, Herning
  - Hvidovre Hospital, Hvidovre
  - Lille Baelt Hospital, Kolding
  - Slagelse Sygehus, Slagelse
- CRC-Alexandria University, Alexandria, Egypt
- Finland (9):
  - CRST Helsinki Oy, Helsinki
  - Terveystalo Ruoholahti, Helsinki
  - Helsinki yliopistollinen sairaala, Helsinki
  - StudyCor Oy, Jyväskylä
  - Itä-Suomen yliopisto/Health Step Finland Oy, Kuopio
  - Suomen Terveystalo oy Tampere, Tampere
  - Tampere University Hospital, Tampere
  - Turun Yliopistollinen sairaala, Turku
  - Terveystalo Pulssi, Turku, Turku
- France (42):
  - HOP de Mercy, Ars-Laquenexy
  - HOP Jean Minjoz, Besançon
  - HOP Ambroise Paré, Boulogne-Billancourt
  - HOP de la Cavale Blanche, Brest
  - HOP Louis Pradel, Bron
  - HOP CHU Caen, Caen
  - HOP William Morey, Chalon-sur-Saône
  - HOP Chambéry, Chambéry
  - HOP Trousseau, Chambray-lès-Tours
  - HOP Sud Francilien, Corbeil-Essonnes
  - Centre Cardiologique d'Evecquemont, Évecquemont
  - Groupe hospitalier mutualiste de Grenoble, Grenoble
  - HOP Haguenau, Haguenau
  - HOP Est Francilien, Jossigny
  - HOP la Rochelle Ré Aunis, La Rochelle
  - HOP CHU de Grenoble, La Tronche
  - HOP André Mignot, Le Chesnay
  - HOP Louis Pasteur, Le Coudray
  - INS Coeur Poumon, Lille
  - HOP Saint Joseph Saint Luc, Lyon
  - HOP Saint Joseph Marseille, Marseille
  - HOP Nord, Marseille
  - HOP Est Francilien Meaux, Meaux
  - Clinique du Millénaire, Montpellier
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pasteur, Nice
  - HOP Lariboisière, Paris
  - HOP La Pitié Salpêtrière, Paris
  - HOP Européen G. Pompidou, Paris
  - HOP Bichat, Paris
  - HOP Pau, Pau
  - HOP Haut-Lévêque, Pessac
  - HOP la Milétrie, Poitiers
  - HOP Cornouaille, Quimper
  - HOP Maison Blanche, Reims
  - HOP Saint-Brieuc, Saint-Brieuc
  - HOP Nord Laennec, Saint-Herblain
  - HOP Civil, Strasbourg
  - Hôpital Rangueil - CHU de Toulouse, Toulouse
  - HOP de Troyes, Troyes
  - HOP Brabois, Vandœuvre-lès-Nancy
  - GH Les Portes du Sud, Vénissieux
- Germany (89):
  - Zentrum für Klinische Studien Bad Homburg, Bad Homburg
  - Universitätsklinikum Freiburg, Bad Krozingen
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, Bad Oeynhausen
  - Kardiologie im Spreebogen, Berlin
  - FutureMeds GmbH, Berlin
  - Velocity Clinical Research Germany GmbH, Berlin, Berlin
  - Policum Berlin Studien GmbH, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - KARDIA - Dr. Hashemi, Berlin
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil gGmbH, Bochum
  - Diabetes- und Stoffwechselpraxis Bochum, Bochum
  - Kardiologisch-Angiologische Praxis, Bremen
  - RKH Fürst-Stirum-Klinik Bruchsal, Bruchsal
  - SANA Kliniken Oberfranken Coburg GmbH, Coburg
  - Gemeinschaftspraxis Kardiologie Köln, Cologne
  - MVZ Dachau Verbund, Dachau
  - Kardiovaskuläres Zentrum Darmstadt, Darmstadt
  - St. Johannes Hospital Dortmund, Dortmund
  - Facharztzentrum Dresden-Neustadt Betriebsgesellschaft mbH, Dresden
  - Herzzentrum Dresden GmbH Universitaetsklinik, Dresden
  - Technische Universität Dresden, Dresden
  - StudyPoint Duisburg GbR, Duisburg
  - Deutsches Diabetes Zentrum DDZ, Düsseldorf, Düsseldorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Diabetologie, Angiologie & Innere Medizin, Eisenach
  - Katholisches Kranken-haus "St. Johann Nepomuk", Erfurt
  - InnoDiab Forschung GmbH, Essen
  - Elisabeth-Krankenhaus Essen GmbH, Essen
  - Klinisches Forschungszentrum Dr. Hagemann, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Gemeinschaftspraxis Denger & Pfitzner, Friedrichsthal
  - Asklepios Harzkliniken GmbH, Goslar
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Diabetes Zentrum Wilhelmsburg GbR, Hamburg
  - Velocity Clinical Research Germany GmbH Hamburg, Hamburg
  - Kardiologie Haßloch, Haßloch
  - St. Elisabeth Gruppe GmbH Katholische Kliniken Rhein-Ruhr, Herne
  - Universität des Saarlandes, Homburg
  - Praxisgemeinschaft Jerichow, Jerichow
  - Kardiopraxis Schirmer, Kaiserslautern
  - B. Braun Ambulantes Herzzentrum Kassel MVZ GmbH, Kassel
  - Zentrum für Klinische Forschung Köln, Köln-Dünnwald
  - Velocity Clinical Research Germany GmbH, Leipzig, Leipzig
  - Familienmedizinisches Zentrum Radowsky, Leipzig
  - Helios Herzzentrum Leipzig GmbH, Leipzig
  - Sana Klinikum Lichtenberg, Lichtenberg
  - Cardio Centrum Ludwigsburg Bietigheim CCLB, Ludwigsburg
  - Kardiologische Praxis Ludwigshafen, Ludwigshafen am Rhein
  - Praxis Oedeme, Lüneburg
  - Institut für Präventive Medizin und Klinische Forschung GbR Prof. Möricke, Magdeburg
  - Cardiopraxis Mainz Ingelheim, Mainz
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - PSHI Praxis GmbH, Mainz
  - ze:ro Praxen MVZ fuer Nierenerkrankungen und Bluthochdruck GmbH Mannheim, Mannheim
  - Praxis Dr. Jens Taggeselle, Markkleeberg
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Gemeinschaftspraxis Dr.med. Martin Prohaska und Dr. med. Felix Schulte, Mühldorf
  - CDG-Zentrum für Diagnostik und Gesundheit, München
  - Institut für Diabetesforschung Münster GmbH, Münster
  - Praxis Dr. Schriek und Kollegen, Münster
  - Marienhaus Klinikum St. Elisabeth, Neuwied
  - Rahman & Detho Studien GmbH, Obertshausen
  - FutureMeds GmbH, Offenbach
  - R.E.D. Institut fuer medizinische Studien und Fortbildung GmbH, Oldenburg in Holstein
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Kardiologische Praxis Papenburg, Papenburg
  - Kardiologische Gemeinschaftspraxis Dres. med. Martin Fleckenstein/Nicola Eberl/Tilmann Pohl/Moritz Rumpf, Penzberg
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam
  - Praxis Reinfeld Mitte, Reinfeld
  - Medizinisches Versorgungszentrum Riesa am Klinikum Döbeln GmbH, Riesa
  - Rostock University Medical Center, Rostock
  - Nephrologische Gemeinschaftspraxis, Hamann/Bacinovic/Jacobsen, Rotenburg (Wümme)
  - Gesundheitsverbund Landkreis Konstanz gGmbH, Singen
  - Barmherzige Brueder gemeinnuetzige Traeger GmbH, Straubing
  - Kardiologische Praxis im Steiner Thor, Straubing
  - Praxisgemeinschaft Melcherstätte, Stuhr
  - Robert Bosch Gesellschaft für medizinische Forschung mbH, Stuttgart
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Praxis Dr. med. Astrid Schmidt-Reinwald, Trier
  - Universitätsklinikum Ulm, Ulm
  - Cardiologicum Hamburg GbR, Wandsbek
  - Zentrum für Klinische Forschung Wangen, Wangen
  - Josephs-Hospital Warendorf, Warendorf
  - Medislim GmbH, Weinheim
  - Kardiologische Praxis, Wermsdorf, Wermsdorf
  - Evangelisches Krankenhaus Witten, Witten
  - Klinikum Worms gGmbH, Worms
  - Praxis für Innere Medizin, Zwenkau
  - Heinrich Braun Klinikum gemeinnützige GmbH, Zwickau
- Greece (16):
  - Evangelismos Hospital of Athens, Athens
  - General Hospital of Athens "Laiko", Athens
  - University Hospital of Athens, Athens
  - Chest Hospital of Athens "Sotiria", Athens
  - General Hospital of Athens "Alexandra", Athens
  - University General Hospital Attikon, Chaïdári
  - General Hospital Venizeleio, Heraklion
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - General University Hospital of Larissa, Larissa
  - Athens Medical Group, Psychikó
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
  - Aristotle University, Thessaloniki, Thessaloniki
  - General Hospital G. Gennimatas, Thessaloniki
  - Nexthealth S.A, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
  - Hospital of Heraklion (PAGNI), Voútai
- Hong Kong (4):
  - Queen Elizabeth Hospital-Hong Kong-51727, Hong Kong
  - Gleneagles Hospital Hong Kong, Hong Kong
  - Prince of Wales Hospital-Hong Kong-20715, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (15):
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - Pericardio Kft., Békéscsaba
  - Belvaros-Lipotvaros Egeszsegugyi Szolgalat, Budapest
  - Geomedical Kft., Budapest
  - Gottsegen National Cardiovascular Center, Budapest
  - Bajcsy-Zsilinszky Hospital and Clinic, Budapest
  - Semmelweis University, Faculty of Medicine, Budapest
  - Privat Doktor SMO, Budapest
  - Central Hospital of Northern Pest - Military Hospital, Budapest
  - BKS Research Ltd, Hatvan
  - Somogy County Kaposi Mor Teaching Hospital, Kaposvár
  - Selye Janos Hospital Komarom, Komárom
  - Coromed-Smo Kft., Pécs
  - University of Pecs, Pécs
  - Tolna County Balassa Janos Hospital, Szekszárd
- India (18):
  - Gujarat Endocrine Centre, Ahmedabad
  - Bangalore Medical College, Bengaluru
  - SP medical college and associated group of hospitals, Bikaner
  - G S V M, Kanpur, Kanpur
  - Apollo Multispeciality Hospitals Limited, Kolkata
  - Rabindranath Tagore International Institute of Cardiac Sciences, Kolkata
  - Kamal Nayan Bajaj Hospital, Maharashtra
  - Diabetes Care and Research Centre, Nagpur
  - Chopda Medicare and Research Centre Pvt Ltd, Nashik
  - GB Pant Hospital, New Dehi
  - Fortis Hospital, New Delhi
  - Sir Gangaram Hospital, New Delhi
  - Batra Hospital and Medical Research Centre, New Delhi
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Max Super Specialty Hospital, Saket, Saket
  - Nirmal Hospital, Surat
  - Jothydev's Diabetes Research Centre, Trivandrum
  - King George Hospital, Visakhapatnam
- Ireland (3):
  - Portiuncula University Hospital, Ballinasloe
  - Connolly Hospital Blanchardstown, Dublin
  - University Hospital Galway, Galway
- Israel (15):
  - Haemek Medical Center, Afula
  - Assuta Medical Center, Ashdod
  - Barzilai Medical Center, Ashkelon
  - Lady Davis Carmel Medical Center, Haifa
  - Linn Medical Center, Haifa
  - Diabetes Institute Herzliya, Herzelia
  - Wolfson Medical Center, Holon
  - Clalit Cardio Community, Holon
  - Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center Beilinson, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
  - Diabetes Medical Center, Tel Aviv
- Italy (28):
  - Ospedale Generale Regionale 'F. Miulli", Acquaviva Delle Fonti (BA)
  - ASST Papa Giovanni XXIII, Bergamo
  - ARNAS Garibaldi Di Catania, Catania
  - Università degli Studi "Magna Grecia", Catanzaro
  - Azienda Sanitaria Locale 2 Lanciano Vasto Chieti, Chieti
  - University Hospital Of Ferrara, Cona (FE)
  - Azienda Sanitaria Locale Avezzano Sulmona L'Aquila, Coppito (AQ)
  - Azienda Ospedaliera-Universitaria Di Cosenza ("SS. Annunziata"), Cosenza
  - A. O. Universitaria Careggi, Florence
  - IRCCS MultiMedica, Milan
  - Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele S.r.l., Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - ARNAS Civico, Palermo
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda Sanitaria Locale TO3, Rivoli (TO)
  - A.O. San Camillo Forlanini, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Azienda Sociosanitaria Ligure 2, Savona
  - Azienda Ospedaliera Universitaria Citta Della Salute E Della Scienza Di Torino, Torino
  - Azienda Ospedaliero Universitaria delle Marche, Torrette (AN)
  - ASST dei Sette Laghi, Tradate (VA)
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
  - ASST dei Sette Laghi, Varese
- Japan (80):
  - Kariya Toyota General Hospital, Aichi, Kariya
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - Japan Community Healthcare Organization Chukyo Hospital, Aichi, Nagoya
  - Nagoya University Hospital, Aichi, Nagoya
  - Chiba University Hospital, Chiba, Chiba
  - Japan Institute for Health Security National Kohnodai Medical Center, Chiba, Ichikawa
  - Chibanishi General Hospital, Chiba, Matsudo
  - Chibaken Saiseikai Narashino Hospital, Chiba, Narashino
  - Ehime Prefectural Central Hospital, Ehime, Matsuyama
  - Saiseikai Matsuyama Hospital, Ehime, Matsuyama
  - Fukuokaken Saiseikai Futsukaichi Hospital, Fukuoka, Chikushino
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Japanese Red Cross Fukuoka Hospital, Fukuoka, Fukuoka
  - Japanese Red Cross Maebashi Hospital, Gumma, Maebashi
  - Gunma Saiseikai Maebashi Hospital, Gumma, Maebashi
  - National Hospital Organization Takasaki General Medical Center, Gumma, Takasaki
  - Hiroshima Red Cross Hospital and Atomic-bomb Survivors Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Hiroshima, Kure
  - Kure Kyosai Hospital, Hiroshima, Kure
  - Asahikawa Medical University Hospital, Hokkaido, Asahikawa
  - Teine Keijinkai Hospital, Hokkaido, Sapporo
  - Manda Memorial Hospital Diabetes Center, Hokkaido, Sapporo
  - Hanaoka Seishu Memorial Hospital, Hokkaido, Sapporo
  - Nishinomiya Watanabe Cardiovascular Cerebral Center, Hyogo, Nishinomiya
  - Hyogo Prefectural Nishinomiya Hospital, Hyogo, Nishinomiya
  - NHO Mito Medical Center, Ibaraki, Higashiibaraki-gun
  - Iryouhouijneiwakai Minamiakatsuka Clinic, Ibaraki, Mito
  - Naka Memorial Clinic, Ibaraki, Naka
  - Tsukuba Medical Center Hospital, Ibaraki, Tsukuba
  - Kanazawa University Hospital, Ishikawa, Kanazawa
  - National Hospital Organization Kanazawa Medical Center, Ishikawa, Kanazawa
  - Iwate Prefectural Central Hospital, Iwate, Morioka
  - Mitoyo General Hospital, Kagawa, Kanonji
  - Kagawa Prefectural Central Hospital, Kagawa, Takamatsu
  - Yokoi Medical Clinic, Kagawa, Takamatsu
  - Tenyoukai Central Clinic, Kagoshima, Kagoshima
  - Nanpuh Hospital, Kagoshima, Kagoshima
  - Tokushukai Hayama Heart Center, Kanagawa, Miura-gun
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Yokohama Rosai Hospital, Kanagawa, Yokohama
  - Yokohama City University Hospital, Kanagawa, Yokohama
  - Yokohama Minami Kyousai Hospital, Kanagawa, Yokohama
  - Chikamori Hospital, Kochi, Kochi
  - Kumamoto University Hospital, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Kyoto Medical Center, Kyoto, Kyoto
  - Tohoku Kosai Hospital, Miyagi, Sendai
  - Sendai Cardiovascular Center, Miyagi, Sendai
  - Shinden Higashi Clinic, Miyagi, Sendai
  - Medicalcity East Hospital, Miyazaki, Miyakonojo
  - Shinshu University Hospital, Nagano, Matsumoto
  - Nagasaki Harbor Medical Center, Nagasaki, Nagasaki
  - Juzenkai The Sakakibara Heart Institute of Okayama, Okayama, Okayama
  - Okayama City General Medical Center Okayama City Hospital, Okayama, Okayama
  - Okayama Rosai Hospital, Okayama, Okayama
  - Nozaki Tokushukai Hospital, Osaka, Daito
  - Matsubara Tokushukai Hospital, Osaka, Matsubara
  - Matsushita Memorial Hospital, Osaka, Moriguchi
  - Ikebuchi Clinic, Osaka, Osaka
  - Chibune General Hospital, Osaka, Osaka
  - National Cerebral and Cardiovascular Center, Osaka, Suita
  - Saiseikai Senri Hospital, Osaka, Suita
  - Ageo Central General Hospital, Saitama, Ageo
  - Koshigaya Municipal Hospital, Saitama, Koshigaya
  - San-Ai Hospital, Saitama, Saitama
  - Saino Clinic, Saitama, Tokorozawa
  - Fujieda Municipal General Hospital, Shizuoka, Fujieda
  - Shizuoka Medical Center, Shizuoka, Sunto-gun
  - Dokkyo Medical University Hospital, Tochigi, Shimotsuga-gun
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Tokushima University Hospital, Tokushima, Tokushima
  - Minamino Cardiovascular Hospital, Tokyo, Hachioji
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
  - Toranomon Hospital, Tokyo, Minato-ku
  - Tokyo Saiseikai Central Hospital, Tokyo, Minato-ku
  - Tokyo Rosai Hospital, Tokyo, Ota-ku
  - Toyama Prefectural Central Hospital, Toyama, Toyama
  - Fujita Health University Hospital, Toyoake-shi
- Latvia (8):
  - Daugavpils Regional Hospital LTD Centre Outpatient Clinic, Daugavpils
  - Zemgale Diabetes Centre, Jelgava
  - Lijas Moras Medical Practice Ltd, Ogre
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East University Hospital, Riga
  - Professor Skride's Heart Clinic, LLC., Riga
  - Sigulda Hospital, Sigulda
  - Gita Rancane's private cardiologist practice, LLC., Ventspils
- Lithuania (7):
  - JSC Klinikiniai sprendimai, Alytus
  - JSC Klinikiniai sprendimai, Kaunas
  - Saules Family Medical Centre, Kaunas
  - Inmedica, Kaunas
  - Klaipeda university hospital, Klaipėda
  - JSC Inlita, Vilnius
  - Vilnius University Hospital, Santariskiu, Vilnius
- Malaysia (10):
  - Hospital Pulau Pinang, George Town
  - Hospital Raja Perempuan Zainab II, Kelantan
  - Sarawak Heart Centre, Kota Samarahan
  - Institut Jantung Negara, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Sarawak General Hospital, Kuching
  - Hospital Miri, Miri
  - Hospital Universiti Teknologi MARA, Sungai Buloh, Sungai Buloh
- Mexico (18):
  - Medical Center Metas S.C., Chihuahua City
  - Instituto de Diabetes, Obesidad y Nutrición S.C., Cuernavaca
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C., Culiacán
  - Instituto Jalisciense de Investigacion En Diabetes Y Obesidad Sc, Guadalajara
  - Virgen Cardiovascular Research SC., Guadalajara
  - Clinica Omega Diabetes, Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Köhler & Milstein Research S.A. de C.V., Mérida
  - Medical Care and Research, Mérida
  - Centro Mexicano de Desarrollo de Estudios Clínicos SA -CEMDEC, México
  - Clinstile S.A. de C.V., México
  - CEINV Salud, S.A. de C.V., Monterrey
  - Cardiolink Clin Trials S.C., Monterrey
  - Unidad Biomédica Avanzada Monterrey, Monterrey
  - Centro Medico Zambrano Hellion, Monterrey
  - Centro de Investigación y Control Metabólico, S.C., Monterrey
  - CIMAB S.A. de C.V., Torreón
  - Sociedad de Metabolismo y Corazón S.C., Veracruz
- Netherlands (24):
  - Jeroen Bosch Ziekenhuis-Hertogenbosch, 's-Hertogenbosch
  - Progress Clinical Research Den Bosch, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
  - Progress Clinical Research Amsterdam, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Amsterdam UMC Locatie AMC, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Rode Kruis Ziekenhuis, Beverwijk
  - PT & R, Born
  - Reinier de Graaf Gasthuis, Delft
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - TREANT zorggroep, Emmen
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Universitair Medisch Centrum Groningen, Groningen
  - Tergooi Ziekenhuis, Hilversum
  - Maastricht University Medisch Centrum, Maastricht
  - Radboud Universitair Medisch Centrum, Nijmegen
  - D&A Research and Genetics, Sneek
  - Diakonessenhuis Utrecht, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medical Center, Venlo
  - Isala Zwolle, Zwolle
  - Progress Clinical Research Zwolle, Zwolle
- New Zealand (5):
  - Christchurch Heart Institute, Christchurch, Canterbury
  - Hutt Hospital, Lower Hutt, Wellington Region
  - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Grafton / Auckland
  - North Shore Hospital, Takpuna Auckland
- Norway (11):
  - Sørlandet sykehus HF, Avd. Arendal, Arendal
  - Nordlandssykehuset HF, Bodø, Bodø
  - Vestre Viken HF, Drammen Sykehus, Drammen
  - Sykehuset Østfold HF, avd. Kalnes, Grålum
  - Akershus Universitetssykehus HF, Lørenskog
  - Colosseumklinikken Dr. Gullestad, Oslo
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
  - Oslo Universitetssykehus HF, Ullevål sykehus, Oslo
  - Skedsmo Medisinske Senter, Skedsmokorset
  - Helse Stavanger, Stavanger Universitetssykehus, Stavanger
  - St. Olavs Hospital, Universitetssykehuset i Trondheim, Trondheim
- Philippines (9):
  - St. Lukes Medical Center Global City, City of Taguig
  - CARE Clinical Trial Group, Dasmariñas
  - Davao Doctors Hospital, Davao City
  - Mary Mediatrix Medical Center, Lipa City
  - Manila Med Medical Centre Manila, Manila
  - Institute for Studies on Diabetes Foundation Inc., Marikina City
  - The Medical City, Pasig
  - St. Luke's Medical Center-Quezon-59457, Quezon City
  - Cardinal Santos Medical Center, San Juan City
- Poland (28):
  - Celenus Sp. z o.o. sp.k., Bełchatów
  - Medical University of Bialystok, Bialystok
  - Centrum Medyczne "Hipokrates" S.C. Elżbieta I Grzegorz Grześk, Bydgoszcz
  - Pratia S.A., Bydgoszcz
  - Pratia S.A., Chojnice
  - Pratia S.A., Częstochowa
  - Clinical Research Center Mital Site, Elblag
  - Pratia S.A., Gdynia
  - FutureMeds Sp. z o.o., Gdynia
  - Pro Familia Altera Sp. z o.o., Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Salvia Lekston I Madej Sp. J., Katowice
  - FutureMeds Sp. z o.o., Krakow
  - Pro Salus Sp. z o.o. sp.k., Lodz
  - Med-Gastr Medical Center, Lodz
  - FutureMeds Sp. z o.o., Lodz
  - Polish Mother's Memorial Hospital - Research Institute, Lodz
  - FutureMeds Sp. z o.o., Olsztyn
  - University Clinical Hospital in Opole, Opole
  - Velocity Nova Sp z o.o., Staszów
  - FutureMeds Sp. z o.o., Warsaw
  - Prof. W. Orlowski Independent Public Clinical Hospital, Warsaw
  - Balsammedica Sp. z o. o., Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - National Geriatrics, Rheumatology and Rehabilitation Institute, Warsaw
  - Royalderm Sp. z o.o., Warsaw
  - FutureMeds Sp. z o.o., Warszawa-Targówek
  - FutureMeds Sp. z o.o., Wroclaw
- Portugal (20):
  - ULS de Almada -Seixal, E. P. E. - Hospital Garcia de Orta, Almada
  - ULS de Amadora/ Sintra, E.P.E. - Hospital Professor Doutor Fernando Fonseca, Amadora
  - ULS da Região de Aveiro, Aveiro
  - ULS Braga, Braga
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Casa de Saúde Santa Filomena, Coimbra
  - ULS do Alto Ave, Guimarães
  - Hospital São Francisco, Leiria
  - Hospital de Santa Marta, Lisbon
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - ULS de Lisboa Ocidental, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital Cruz Vermelha, Lisbon
  - ULS de Santa Maria, E.P.E, Lisbon
  - Unidade Local de Saúde de Matosinhos, Matosinhos Municipality
  - Centro Hospitalar Universitário São João,EPE, Porto
  - ULS de Entre Douro e Vouga, Santa Maria da Feira
  - ULS do Estuário do Tejo, Vila Franca de Xira
  - Hospital da Luz Arrábida, Vila Nova de Gaia
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E, Vila Nova de Gaia
- Puerto Rico (6):
  - Dorado Medical Complex, Dorado
  - Ponce School of Medicine/CAIMED Center, Ponce
  - Research and Cardiovascular Corporation, Ponce
  - Latin Clinical Trial Center, San Juan
  - GCM Medical Group, PSC, San Juan
  - FDI Clinical Research, San Juan
- Romania (24):
  - S.C. Diana Barbonta S.R.L, Alba Iulia
  - Individual Medical Practice Dr. Mercea Corina Delia, Baia Mare
  - Individual Medical Practice Dr. Calin Pop, Baia Mare
  - Spitalul Judetean de Urgenta Braila, Brăila
  - Clinica Medicala Data Plus SRL, Bucharest
  - SC Nicodiab SRL, Bucharest
  - Hightech Medical Services, Bucharest
  - National Institute of Diabetes, Nutrition, Metabolic Diseases Prof. Dr. N.Paulescu, Bucharest
  - Institutul de Urgenta pentru Boli Cardiovasculare "Prof.Dr.C.C.Iliescu", Bucharest
  - Emergency University Hospital, Bucharest
  - Societatea Civila Medicala Dr. Paveliu, Bucharest
  - Mat Cord Biomedica S.R.L., Buzău
  - Milena Sante, Galati
  - Diamed Obesity SRL, Galati
  - Consultmed SRL, Iași
  - SC Cardiomed SRL, Iasi, Iași
  - Diabdana S.R.L., Oradea
  - Sal Med Srl, Piteşti
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - Mediab S.R.L., Târgu Mureş
  - Podoleanu G. Cristian-Gheorghe-Calin, Târgu Mureş
  - Fundatia Cardioprevent, Timișoara
  - Cabinet Medical Dr. Geru SRL, Timișoara
  - S.C Medicali's S.R.L, Timișoara
- Saudi Arabia (6):
  - Imam Abdulrahman bin Faisal University, Dammam
  - King AbdulAziz University Hospital, Jeddah
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - King Fahad Medical City, Riyadh
  - King Saud Medical City, Riyadh
  - Al Habib Medical Group, Riyadh
- Serbia (7):
  - Clinical Hospital Center Dr. Dragisa Misovic, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - University Clinical Center of Kragujevac, Kragujevac
  - Institute for Treatment and Rehabilitation, Niska Banja, Niška Banja
  - General Hospital Pancevo, Pančevo
  - Institute of Cardiovascular Diseases of Vojvodine, Sremska Mitrovica
- Singapore (5):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
- Slovakia (8):
  - Kardiointerna s r o, Banská Bystrica
  - Alian s.r.o., Bardejov
  - Premedix Clinic, Bratislava
  - Vysokospecializovany Odborny ustav Geriatricky sv. Lukasa v Kosiciach n.o., Košice
  - MEDI M&M, Moldava nad Bodvou
  - Dentavia s.r.o., Poprad
  - Interna SK, Svidník
  - JAL s.r.o., Trnava
- South Africa (28):
  - Lakeview Hospital, Benoni
  - Iatros International, Bloemfontein
  - TREAD Research, Cape Town
  - Langeberg Clinical Trials, Cape Town
  - Paarl Research Centre, Cape Town
  - Johese Clinical Research: Midstream, Centurion Gauteng
  - Canal Walk Clinical Trial Centre, Century City
  - Prof N Ranjith Cardiovascular Research Centre, Durban
  - Synapta Clinical Research Centre, Durban
  - Clinresco Centre, Gauteng
  - Diabetes Care Centre, Johannesburg
  - Life The Glynnwood, Johannesburg
  - Drs H & V Makan, Johannesburg
  - Lenasia Clinical Trial Centre, Johannesburg
  - Dr Garda Cardiology Practice, Johannesburg
  - Meditrial, Pietermaritzburg
  - Dr I.O Ebrahim Inc, Pretoria
  - Diabetes Care Centre, Pretoria
  - Jongaie Research, Pretoria
  - Clinical Trial Systems (Pty) Ltd, Pretoria
  - Global Clinical Trials, Raslouw
  - Helderberg Research Institute, Somerset West
  - Vergelegen Medi-Clinic, Somerset West
  - Wits Clinical Research Chris Hani Baragwanath Hospital, Soweto
  - Tiervlei Trial Centre, Tygervalley
  - Tickerdoc Research (Pty) LTD, West Wing
  - Clinical Projects Research, Worcester
  - CareKahle Pty Ltd, Wynberg
- South Korea (17):
  - Korea University Ansan Hospital, Ansan-si
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Eulji University Hospital, Daejeon
  - Chungnam National University Hospital, Daejoen
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (21):
  - Hospital Germans Trias i Pujol, Badalona
  - Centro Médico Teknon, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves, Beiro
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital de Galdakao, Galdakao
  - Hospital Infanta Elena, Huelva
  - Hospital Universitario de Jaén, Jaén
  - Hospital de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - CS Parc Taulí, Sabadell
  - Centro Atención Primaria La Mina, Sant Adrià de Besòs
  - Hospital Universitario Marqués de Valdecilla, Santader
  - Hospital Virgen del Rocío, Seville
  - Hospital General Universitario de Toledo, Toledo
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Río Hortega Valladolid, Valladolid
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital Virgen de las Montañas, Villamartín
- Sweden (15):
  - Södra Älvsborgs Sjukhus, Borås
  - Falu lasarette, Falun
  - Forskningsenheten Carlanderska, Gothenburg
  - Sahlgrenska Universitetssjukhuset, Östra, Gothenburg
  - Hallands sjukhus Halmstad, Halmstad
  - Centralsjukhuset Karlstad, Karlstad
  - Lasarettet Ljungby, Ljungby
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Södertälje Sjukhus, Södertälje
  - Capio St. Görans Sjukhus, Stockholm
  - Akademiskt Specialistcentrum Centrum för Diabetes, Stockholm
  - Danderyds Sjukhus, Stockholm
  - Länssjukhuset Sundsvall Härnösand, Sundsvall
  - Norrlands universitetssjukhus, Umeå
  - Centrallasarettet Växjö, Vaxjo
- Switzerland (6):
  - Universitätsspital Basel, Basel
  - University Hospital of Lausanne, Lausanne
  - Lucerne Cantonale Hospital, Lucerne
  - Cantonal Hospital Organization - Ente Ospedaliero Cantonale (EOC), Lugano
  - HOCH Health Ostschweiz, Sankt Gallen
  - University Hospital Zurich, Zurich
- Taiwan (13):
  - Chia-Yi Christian Hospital, Chia-Yi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Thailand (10):
  - Vajira Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiangmai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - Naresuan University Hospital, Phitsanulok
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (20):
  - Adana City Hospital, Adana
  - Baskent University Hospital, Adana
  - Afyonkarahisar Health Sciences University Hospital, Afyonkarahisar
  - University of Health Sciences, Ankara Gulhane Training and Research Hospital, Ankara
  - Ankara Üniversitesi İbn-i Sina Hastanesi, Ankara
  - Gazi University Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Bursa Uludag University, Bursa
  - Bursa Şehir Hastanesi, Bursa
  - Trakya University Hospital, Edirne
  - İstanbul Çapa University, Istanbul
  - İstanbul Prof.Dr. Cemil Taşçıoğlu City Hospital, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Göztepe City Hospital, Istanbul
  - Dokuz Eylul University Faculty of Medicine, Izmir
  - Erciyes University, Kayseri
  - Inonu University Turgut Ozal Medical Center, Malatya
  - Siyami Ersek Heart Hospital, Uskudar / Istanbul
  - Zonguldak Bulent Ecevit University, Obesity and Diabetes Research and Application Center, Zonguldak
- United Kingdom (33):
  - FutureMeds - Birmingham, Birmingham
  - Royal Blackburn Teaching Hospital, Blackburn
  - Glan Clwyd Hospital, Bodelwyddan
  - Royal Bournemouth Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Coniston Medical Practice, Bristol
  - Yatton Surgery, Bristol
  - FutureMeds - Liverpool, Bromborough
  - St Richard's Hospital, Chichester
  - Queen Alexandra Hospital, Cosham
  - Darlington Memorial Hospital, Darlington
  - Royal Derby Hospital, Derby
  - Ninewells Hospital & Medical School, Dundee
  - The Falmouth Health Centre Practice, Falmouth
  - The Garth Surgery, Guisborough
  - Ipswich Hospital (UK), Ipswich
  - Victoria Hospital, Kirkcaldy
  - Royal Lancaster Infirmary, Lancaster
  - Pinfold Surgery, Leeds
  - Lincoln County Hospital, Lincoln
  - William Harvey Research Limited, London
  - FutureMeds - London, London
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital, Manchester
  - North Manchester General Hospital, Manchester
  - Linthorpe Surgery, Middlesbrough
  - Mayford House Surgery, Northallerton
  - Norfolk and Norwich University Hospital, Norwich
  - Moorgreen Hospital, Southampton
  - Swansea University Medical School, Swansea
  - Trowbridge Health Centre, Trowbridge
  - Weymouth Research Hub, Weymouth
  - Woodthorpe Surgery, York
- Vietnam (4):
  - Hanoi Medical University, Hanoi
  - People's Hospital 115, Ho Chi Minh City
  - Thong Nhat Hospital HCMC, Ho Chi Minh City
  - University Medical Center HCMC, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency